CLINICAL TRIAL: NCT06277063
Title: Noninvasive Vagus Nerve Stimulation for the Prevention and Treatment of Primary Headache: a Single-arm Single-center Clinical Trial.
Brief Title: nVNS for the Prevention and Treatment of Primary Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: BrainClos Company, LTD. (Unknown); Zhuhai Fudan Innovation Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-057
Record Dates: First submitted 2024-02-04; First posted 2024-02-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Primary Headache; Migraine in Adolescence; Migraine in Children; Cluster Headache; Tension Headache
Keywords: Primary headache; Adolescents; Noninvasive vagus nerve stimulation
MeSH Terms: conditions — Cluster Headache; Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute exacerbation experimental group (Experimental): VAS pain intensity will be assessed at the onset of headache, and patients will receive nVNS for half an hour within 20 minutes of the onset, and post-treatment evaluation results will be recorded immediately after treatment, 2 hours, 8-12 hours, 24 hours, and 36-48 hours. During the course of treatment and intervention, a 20-minute ECG closed-loop assessment test will be performed before admission and after return. The procedure included: 5 minutes of rest (i.e. no vagal stimulation), 10 minutes of vagal stimulation, 5 minutes of rest(5-10-5), a total of 20 minutes of ECG, and real-time extraction of heart rate and sex data. Neck electromyography before and after intervention was also used as an auxiliary indicator.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation — The vagus nerve's auricular branch is primarily distributed in the tragus, tragus sulcus, and concha cavity. It can activate the nucleus tractus solitarius through the vagus afferent fibers, thereby activating various areas of the vagus nerve in the central nervous system. This stimulation technique involves applying a constant current of around 2-3mA to the epidermal terminals of the ear using an electrode. It aims to regulate the vagus nerve, modulate the autonomic nervous system, release neurotransmitters, improve cerebral blood flow, and alleviate headache symptoms. In the implementation, non-invasive transcutaneous vagus nerve stimulation was performed by having the subject wear a vagus stimulator and adjusting the appropriate stimulation intensity.

SUMMARY:
This study is a single-center, single-arm study. All subjects will receive the same treatment.

Children and adolescents (7-20 years old) with migraine who met the inclusion criteria will be enrolled as subjects in the experimental group, and the changes in headache scores before and after the intervention will be compared. The intervention method is as follows: ictal intervention, in which subjects will be evaluated for headache improvement after a short intervention during an acute exacerbation. By wearing a vagus stimulator, the stimulating electrode will be located in the concha region rich in vagus nerve fiber endings, and the appropriate stimulation intensity will be adjusted for stimulation.

Therefore, this study will verify the effect of nVNS on the acute treatment of primary headache in children and adolescents. Based on the electrocardiogram and electromyography indicators during the intervention process of nVNS, an objective evaluation system for the improvement of headache by nVNS is established, and the role of stimulation parameters on the effect is further explored to realize the optimization of parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with migraine, cluster headache and tension-type headache were diagnosed according to Chinese Guidelines for the diagnosis and Treatment of Migraine (2022 edition) and Chinese Guidelines for the diagnosis and treatment of cluster headache (2022 edition).
2. Age >=7 years old, <=20 years old;
3. Patients have experienced headache on 3-15 days per month in the past;
4. Maintain a stable dose and frequency of medication and do not take new drugs during the course of participating in the trial;
5. They volunteered to participate in the trial and signed informed consent.

Exclusion Criteria:

1. History of secondary headache, aneurysm, intracranial hemorrhage, brain tumor, severe head trauma, drug abuse, addiction, syncope, or seizures;
2. prior migraine-preventive surgery, cervical vagotomy, or implantation of an electronic or neurostimulator device;
3. Simultaneous use of other devices (e.g., TENS devices, muscle stimulators);
4. An implantable medical device in use, such as a pacemaker, hearing aid, or any implantable electronic device;
5. underwent head and neck nerve block within the past 2 months;
6. Opioid use (more than 2 days per month); Use of analgesics alone or non-steroidal anti-inflammatory drugs (more than 15 days per month); Or tamoxifen, ergots or combination analgesics (more than 10 days per month);
7. Patients who underwent cervical vagotomy (cervical vagotomy);
8. Pediatric patients (under 6 years old); Pregnant women;
9. Patients with clinically significant hypertension, hypotension, bradycardia or tachycardia;
10. Patients with congenital heart disease;
11. Mental/cognitive disorders, etc.

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in pain intensity--actue period study | 2 hours after treatment
  The visual analogue scale (VAS) was used to evaluate the pain. It is widely used in clinical practice in China. The basic method is to use a swimming ruler of about 10cm in length, marked with 10 scales on one side, and "0" and "10" scales on both ends.
  For the AP study, the primary outcome measure is the reduction in pain intensity assessed by VAS 2 hours after treatment.

SECONDARY OUTCOMES:
Heart rate variability(HRV)--actue period study and preventive period study | before and after the intervention. The test consisted of 5 mins of rest (i.e., no vagal stimulation), 10 mins of vagal stimulation, 5 mins of rest, and a total of 20 minutes of electrocard
  A 20-minute closed-loop ECG assessment test was performed before and after the intervention for both the AP study and PP study. The test consisted of 5 minutes of rest (i.e., no vagal stimulation), 10 minutes of vagal stimulation, 5 minutes of rest, and a total of 20 minutes of electrocard.
Electromyography(EMG)--actue period study and preventive period study | before and after the intervention. The test consisted of 5 mins of rest (i.e., no vagal stimulation), 10 mins of vagal stimulation, 5 mins of rest, and a total of 20 minutes of electrocard
  A 20-minute closed-loop evaluation test of neck electromyography was performed before and after the intervention for both the AP study and PP study. The testing process consisted of 5 minutes of rest (i.e., no vagal stimulation), 10 minutes of vagal stimulation, 5 minutes of rest, and a total of 20 minutes of electrocard.
Change in pain intensity--actue period study | half hour, 8-12 hours, 24 hours, and 36-48 hours after treatment
  For the AP study, we will analysis the change in pain intensity assessed by VAS scores, half hour, 8-12 hours, 24 hours, and 36-48 hours after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Ya-Bin, post-doc, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Martelletti P, Barbanti P, Grazzi L, Pierangeli G, Rainero I, Geppetti P, Ambrosini A, Sarchielli P, Tassorelli C, Liebler E, de Tommaso M; PRESTO Study Group. Correction to: Consistent effects of non-invasive vagus nerve stimulation (nVNS) for the acute treatment of migraine: additional findings from the randomized, sham-controlled, double-blind PRESTO trial. J Headache Pain. 2018 Dec 18;19(1):120. doi: 10.1186/s10194-018-0949-9. PMID 30563446
- [Background] Diener HC, Goadsby PJ, Ashina M, Al-Karagholi MA, Sinclair A, Mitsikostas D, Magis D, Pozo-Rosich P, Irimia Sieira P, Lainez MJ, Gaul C, Silver N, Hoffmann J, Marin J, Liebler E, Ferrari MD. Non-invasive vagus nerve stimulation (nVNS) for the preventive treatment of episodic migraine: The multicentre, double-blind, randomised, sham-controlled PREMIUM trial. Cephalalgia. 2019 Oct;39(12):1475-1487. doi: 10.1177/0333102419876920. Epub 2019 Sep 15. PMID 31522546
- [Background] Cao J, Zhang Y, Li H, Yan Z, Liu X, Hou X, Chen W, Hodges S, Kong J, Liu B. Different modulation effects of 1 Hz and 20 Hz transcutaneous auricular vagus nerve stimulation on the functional connectivity of the periaqueductal gray in patients with migraine. J Transl Med. 2021 Aug 17;19(1):354. doi: 10.1186/s12967-021-03024-9. PMID 34404427
- [Background] Lai YH, Huang YC, Huang LT, Chen RM, Chen C. Cervical Noninvasive Vagus Nerve Stimulation for Migraine and Cluster Headache: A Systematic Review and Meta-Analysis. Neuromodulation. 2020 Aug;23(6):721-731. doi: 10.1111/ner.13122. Epub 2020 Mar 12. PMID 32166843
- [Derived] Weng S, Xiao X, Liang S, Xue Y, Yang X, Ji Y. Single-centre, randomised and double-blind clinical trial on the efficacy of transcutaneous auricular vagus nerve stimulation in preventing and treating primary headache in children and adolescents: a study protocol. BMJ Open. 2025 Mar 12;15(3):e092692. doi: 10.1136/bmjopen-2024-092692. PMID 40074270

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Study Protocol (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT06277063/Prot_SAP_ICF_004.pdf
  • Informed Consent Form: Informed Consent Form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT06277063/ICF_005.pdf